CLINICAL TRIAL: NCT03322982
Title: A Randomized, Controlled Trial of Low-fat Diet for Fatigue in Multiple Sclerosis
Brief Title: Low Fat Diet for Fatigue in MS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Vijayshree Yadav, Associate Professor of Neurology, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: OHSU IRB16600
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Multiple Sclerosis
Keywords: diet, low-fat
MeSH Terms: conditions — Multiple Sclerosis | interventions — Diet, Fat-Restricted

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Diet adherence assessments will be conducted by blinded assessors from OHSU bionutrition team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- MS Diet (Experimental): 34 people with MS following low-fat diet
  Interventions: Behavioral: Low-fat diet
- MS Wait-List (No Intervention): 34 people with MS following usual diet
- Diet Healthy Control (No Intervention): 20 controls with no diagnosis of MS, age and sex-matched to members of the MS Diet group
- Wait-List Healthy Control (No Intervention): 20 controls with no diagnosis of MS, age and sex-matched to members of the MS Wait-List group

INTERVENTIONS:
Behavioral: Low-fat diet — less than 20% calories from fat daily
  Arms: MS Diet

SUMMARY:
A randomized, controlled pilot trial of a dietary intervention vs. wait-list control in patients with MS and fatigue for management of their fatigue. The hypothesis of this study is that participants following the low-fat study diet will demonstrate a significant reduction in fatigue after four months compared to wait list controls.

ELIGIBILITY:
For participants with MS:

Inclusion Criteria:

* Age 18-70
* Diagnosis of MS by 2010 McDonald Criteria
* EDSS ≤ 7.5
* Experiencing moderate to severe fatigue (MFIS ≥ 38)

Exclusion Criteria:

* Current cardiopulmonary disease requiring treatment
* Diabetes
* Pregnancy or breast-feeding
* MS exacerbation within 30 days of screening visit
* IV steroids within 30 days of screening visit
* Dietary fat content of <30% as assessed by food frequency questionnaire (FFQ) at screening visit
* Fish oil or flax seed oil supplementation within 30 days of screening visit

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2022-03-31 (Estimated)

PRIMARY OUTCOMES:
Fatigue | Baseline to month 4
  Measured by Modified Fatigue Impact Scale (MFIS). The MFIS is a 21-item questionnaire that assesses overall self-reported fatigue. Subjects rate agreement with a series of statements on a scale of 0 (rarely) to 4 (almost always), in context of their fatigue over the preceding four weeks. Total possible score of 84. Individuals with an MFIS score of > 38 are considered to experience moderate to severe "fatigue

SECONDARY OUTCOMES:
Fatigue | Baseline to month 4
  Measured by Fatigue Severity Scale (FSS). The FSS is a 9-item questionnaire, with subjects giving a response from 1-7 to indicate their degree of agreement with each statement.
Disability | Baseline to month 4
  Measured by EDSS. The EDSS is an eight functional system scale including motor, sensory, cerebellar, brain stem, visual, mental, sphincteric, and other systems. Each functional system is graded from 0 (no disability) to 5 or 6 (maximal disability)20. An integrated score between 0 (normal examination) and 10 (death from MS) is formed based on the score in each functional system.

OTHER OUTCOMES:
Microbiome- Relative abundance of targeted species of gut microflora | Baseline to month 4
  Measured by 16S rRNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Vijayshree Yadav, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chase E, Chen V, Martin K, Lane M, Wooliscroft L, Adams C, Rice J, Silbermann E, Hollen C, Fryman A, Purnell JQ, Vong C, Orban A, Horgan A, Khan A, Srikanth P, Yadav V. A low-fat diet improves fatigue in multiple sclerosis: Results from a randomized controlled trial. Mult Scler. 2023 Nov;29(13):1659-1675. doi: 10.1177/13524585231208330. PMID 37941305